CLINICAL TRIAL: NCT06403475
Title: Transcutaneous Vagus Nerve Stimulation for Language Recovery After Stroke: a Pilot Study
Brief Title: Transcutaneous Vagus Nerve Stimulation in Aphasia After Stroke
Acronym: TRANSLATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STH22935
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Aphasia; Chronic Stroke
Keywords: aphasia; vagus nerve stimulation; stroke; transcutaneous vagus nerve stimulation
MeSH Terms: conditions — Aphasia; Stroke | interventions — Language Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Vagus Nerve Stimulation (Experimental): The intervention will take place for up to 45 minutes per day, 5 days per week for 6 weeks. The stimulation device will be worn whilst completing computer-based Speech and Language Therapy.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation; Behavioral: Computer Based Speech and Language Therapy (Step by Step)
- Sham Transcutaneous Vagus Nerve Stimulation (Sham Comparator): The sham intervention will take place for up to 45 minutes per day, 5 days per week for 6 weeks. The device will be in 'sham' mode. The stimulation device will be worn whilst completing computer-based Speech and Language Therapy.
  Interventions: Device: Sham Transcutaneous Vagus Nerve Stimulation; Behavioral: Computer Based Speech and Language Therapy (Step by Step)

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — Transcutaneous auricular vagus nerve stimulation using the Nurosym (Parasym Ltd) device.
  Stimulation parameters:
  Pulse width: 250µs; Frequency: 25Hz; Intensity: Below pain threshold.
  The active stimulation will be delivered to the left ear. Participants will complete the intervention at home once they have received sufficient training on how to use the stimulation device.
  Arms: Transcutaneous Vagus Nerve Stimulation
Device: Sham Transcutaneous Vagus Nerve Stimulation — Stimulation will be delivered at the same parameters however, sham stimulation will be delivered to the left ear. This sham method has been used as a sham in other studies as it is not thought to activate the vagus nerve.
  Arms: Sham Transcutaneous Vagus Nerve Stimulation
Behavioral: Computer Based Speech and Language Therapy (Step by Step) — Computer-based Speech and Language Therapy will be completed whilst wearing the stimulation device in all groups. The Step by Step programme uses an errorless learning approach to practice naming. All participants will practice a set of 30 meaningful words during the intervention. Participants will complete the SLT programme at home on an ipad, whilst using the stimulation device.

SUMMARY:
Aphasia is an acquired language disorder. Stroke is the most common cause of aphasia, which affects 30% of stroke survivors. Speech and Language Therapy (SLT) can help people with aphasia but it may not be provided at the required intensity. Access to therapy is often limited after the first few months following stroke. People with aphasia can improve with therapy many years after stroke but these benefits have not been found to translate to day to day conversation.

Transcutaneous Vagus Nerve Stimulation (tVNS) is a non-invasive technique which involves stimulating a branch of the vagus nerve through the skin of the ear, using a small earpiece. This technique is safe and has been approved for use in headache. There is promising evidence that tVNS can improve motor rehabilitation in chronic stroke. This technique may be helpful in aiding language recovery in individuals with chronic aphasia.

The current pilot study will primarily assess the feasibility, safety and tolerability of self-directed tVNS paired with computer-based SLT, in individuals with chronic stroke-related aphasia. Secondly, the study aims to explore the effect of the intervention on word-finding ability and to explore potential mechanisms of action. Participants will be randomly allocated to an active or sham tVNS group. Participants will be asked to use the stimulation device at home for 6 weeks, whilst completing computer-based SLT. To date, there are no published studies exploring the use of tVNS in aphasia. An indication of study feasibility may support the development of a larger RCT to explore treatment efficacy.

DETAILED DESCRIPTION:
Aphasia is an acquired communication disorder, characterised by difficulties with the production and/or understanding of language. Stroke is the most common cause of aphasia which affects approximately 30% of stroke survivors. Many individuals are left with chronic deficits. Speech and Language Therapy (SLT) is the gold-standard treatment for aphasia but access to therapy is limited beyond the first few months of recovery. Individuals with chronic aphasia (>6 months) can benefit from SLT input. Computer-based SLT can lead to improvements in word-finding for people with aphasia, many years after stroke (Palmer et al., 2019). Improvements have not been found to translate to day-to-day conversation.

Vagus Nerve Stimulation (VNS) paired with upper limb rehabilitation has proved beneficial in chronic stroke. Transcutaneous Vagus Nerve Stimulation (tVNS) is a non-invasive technique which involves stimulating a branch of the vagus nerve through the skin of the ear, using a small earpiece. This technique is safe and has been approved for use in headache. The use of tVNS in chronic stroke is currently being explored, with promising findings when paired with upper limb rehabilitation exercises. To date, there are no published studies exploring the use of tVNS in chronic aphasia. Pairing tVNS with an SLT intervention may have the potential to promote language recovery in chronic stroke. An indication of study feasibility may support the development of a larger RCT to explore treatment efficacy.

This is a single centre, single blind, pilot randomised controlled trial. The primary aim is to explore the safety, tolerability and feasibility of self-directed computer-based SLT combined with tVNS, in individuals with chronic-stroke related aphasia. Secondary aims include exploring any indication of effect of the intervention on word-finding ability (trained words, generalisability to untrained words and conversation). Additionally, the study aims to explore potential mechanisms of action.

Participants will be asked to use the stimulation device alongside computer-based SLT, at home for 6 weeks. SLT training will include naming pictures of 30 personally relevant words, selected by the participant prior to the commencement of the intervention and uploaded onto the software. The SLT software (Step by Step) uses a self-guided errorless learning approach and will be completed on an ipad. The researcher will check-in with the participant each week to monitor any concerns, side effects and monitor engagement with the programme.

Potential participants will be recruited from Sheffield, using the NHS PHIND database. Accessible study invitations will be sent to potential participants. The Consent Support Tool will be used to ascertain the most appropriate way to provide study information. All participants will have capacity to consent to the study. Participants will be randomly allocated (SealedEnvelope Ltd) to an active or sham tVNS group, stratified according to language score. Participants will be blinded to group allocation.

The tVNS device will be applied to the ear (tragus or earlobe), depending on group allocation. The tVNS device (Nurosym/ Parasym II) is a UKCE marked device, indicated for off-label use in the current study. tVNS use is safe however it has been associated with mild and transitory side effects such as pain or irritation at the stimulation site, headache and nasopharyngitis (Redgrave et al 2018). Stimulation parameters are in line with previous studies:

* Pulse Width: 250µs
* Frequency: 25Hz
* Intensity: individual tolerability (below pain threshold)
* Duration: 45 minutes daily for 6 weeks

Language assessments will be taken at baseline, end of treatment (6 weeks) and at follow-up (12 weeks). To explore potential mechanisms, blood samples, heart rate variability (HRV) and pupillometry measures will be taken at baseline and end of treatment. The Functional near infrared spectroscopy (fNIRS; LUMO, Gowerlabs) will be used on a subset of participants to explore cortical activation in the frontal lobes in response to tVNS at baseline and end of treatment (6 weeks). Outcome measures will be undertaken by a trained member of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial stroke at least 6 months prior to recruitment
* Aphasia (with word finding difficulties)
* Ability to engage in the programme (support can be provided for cognitive or receptive difficulties)
* Sufficient vision to engage in the computer-based SLT programme

Exclusion Criteria:

* Implanted devices (e.g. pacemaker) or implanted stimulation devices
* Currently receiving a programme of Speech and Language Therapy (SLT)
* Damage to the vagus nerve
* Symptomatic bradycardia/ 2nd or 3rd heart block
* Pregnancy
* Unable to speak English
* Severe deafness (despite using hear aids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety: The number of adverse events reported that are associated with tVNS | 6 weeks
  The safety of using tVNS in the aphasia population will be measured through the recording of adverse events. The number of Serious Adverse Events (SAE's) and Unexpected Adverse Events (UAE's) during the intervention will be reported.
Tolerability: The number and intensity of symptoms reported | 6 weeks
  The reporting of symptoms associated with tVNS will be recorded and the severity of each symptom on a 1-5 scale (1= mild; 5 = severe).
Percentage of participants completing the study intervention and outcome measures | 24 months
  >80% of recruited participants completing the intervention and primary outcome measures at 6 weeks

SECONDARY OUTCOMES:
Picture Naming (personally relevant) | Week 0; Week 6; Week 12
  The number of pictures that are accurately named at each time point, out of a maximum of 30. Pictures will be personally relevant and selected by the participant prior to the start of the intervention. These pictures will be trained during the computer-based SLT intervention. Naming will be assessed at baseline, end of treatment (6 weeks) and at follow-up (12 weeks) using the same picture set.
The Comprehensive Aphasia Test (CAT): Naming Objects | Week 0; Week 6; Week 12
  The number of pictures that are accurately named at each time point, out of a maximum of 48. A standardized set of 24 pictures will be used from The Comprehensive Aphasia Test (CAT) Naming Objects subtest. This will assess the ability to name untrained words. This task will be completed at baseline, end of treatment (6 weeks) and at follow-up (12 weeks).
Conversation: The number of trained words used in conversation | Week 0; Week 6; Week 12
  A 10 minute scripted conversation will be conducted for each participant, surrounding topics of personal relevance, to prompt the use of trained words in a conversational context. The number of times a word is used will be recorded
Brain Derived Neurotrophic Factor (BDNF) (ng/ml) | Week 0; Week 6
  Blood samples will be taken at baseline and end of treatment (6 weeks) to measure BDNF levels in serum
Inflammatory markers (pg/ml) | Week 0; Week 6
  Blood samples will be taken at baseline and end of treatment (6 weeks) to measure inflammatory markers: IL-1B, IL-6, IL-10 and TNFa (pg/ml).
Heart Rate Variability (HRV) | Week 0; Week 6
  Heart rate variability will be measured in 5 minute phases before, during and following electrical stimulation. The Standard deviation of the RR intervals (SDNN) will be recorded (ms).
Pupillary Reactivity | Week 0; Week 6
  Pupillary response to light stimulus. Maximum and minimum diameters (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ali Ali, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Prof. Arshad Majid, Study Director — University of Sheffield; Prof. Rebecca Palmer, Study Director — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

REFERENCES:
- [Background] Palmer R, Dimairo M, Cooper C, Enderby P, Brady M, Bowen A, Latimer N, Julious S, Cross E, Alshreef A, Harrison M, Bradley E, Witts H, Chater T. Self-managed, computerised speech and language therapy for patients with chronic aphasia post-stroke compared with usual care or attention control (Big CACTUS): a multicentre, single-blinded, randomised controlled trial. Lancet Neurol. 2019 Sep;18(9):821-833. doi: 10.1016/S1474-4422(19)30192-9. PMID 31397288
- [Background] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648